CLINICAL TRIAL: NCT03918642
Title: Optimizing Psychotherapy for Older Veterans With Chronic Pain
Acronym: OPOVCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURA-013-18F; 1K2CX001884-01A1 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic Pain; Psychotherapy; Musculoskeletal Disease
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Musculoskeletal Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two-Group Parallel Comparison Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emotional Awareness and Expression Therapy (Experimental): Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy
- Cognitive Behavior Therapy (Active Comparator): Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Focus on emotions, writing about stress, assertiveness training, role playing new ways to handle relationships, and sharing feelings and experiences with others.
  Other Names: EAET
  Arms: Emotional Awareness and Expression Therapy
Behavioral: Cognitive Behavior Therapy — Focus on cognitive and behavioral skills, such as relaxation, increasing pleasant activities, pacing, and changing ways of thinking.
  Other Names: CBT
  Arms: Cognitive Behavior Therapy

SUMMARY:
This study is being performed to compare the effects of two alternate types of psychotherapy, Cognitive Behavior Therapy (CBT) and Emotional Awareness and Expression Therapy (EAET), for chronic musculoskeletal pain in older adults. In addition, the investigators will evaluate which patients respond better to each treatment and further investigate how each treatment works. CBT, which focuses on improving coping skills for pain, is the standard form of psychotherapy offered at VA. EAET instead focuses on understanding how life stress, relationships, and emotions may cause and perpetuate pain.

The investigators are performing the study because pain is a large problem among Veterans. Studies show that chronic pain affects as many as 50% of male Veterans and 75% of female Veterans. The investigators are focusing on older adult Veterans because they have the highest rates of chronic pain at VA, perhaps as high as 80%. The investigators are looking at psychotherapy in this study because VA, the Department of Defense, and the CDC recently recommended psychosocial treatments, such as psychotherapy, as first treatments for chronic pain, along with medications other than opioids (e.g., oxycodone). However, only one form of psychotherapy, CBT, is currently available in clinical practice at VA, and this study may provide evidence for making EAET available to Veterans as well.

DETAILED DESCRIPTION:
The overarching goal of the proposed research is to learn how to optimize psychotherapy for those Veterans most in need and most likely to benefit from psychotherapy, older Veterans with chronic musculoskeletal pain. Chronic pain is a critical healthcare challenge, as the condition affects 50% of all Veterans and affects older Veterans most commonly, severely, and persistently. For years, chronic pain treatment has been notoriously difficult at VA and elsewhere, especially in light of the recent "opioid crisis," in which opioid analgesics, previously a mainstay of chronic pain treatment, have come under increased scrutiny. In response, CDC, VA/DoD, and some experts have called for enhancing and expanding psychosocial treatment options for chronic pain, such as psychotherapy, which are low risk for older Veterans who frequently have multiple medical comorbidities and are taking multiple medications.

Yet standard VA psychotherapy approaches, such as Cognitive Behavior Therapy (CBT), have shown modest benefits for Veterans on pain and other related outcomes, such as mood, anxiety, and sleep. In contrast, a novel psychotherapy approach, Emotional Awareness and Expression Therapy (EAET), has shown medium to large benefits for some chronic pain patients. Whereas CBT improves pain and negative emotion by teaching patients cognitive and behavioral coping skills, affecting brain regions that enhance "cognitive control" of pain, EAET operates primarily through emotion regulation, which is thought to influence brain regions and circuits that modulate both physical pain and emotion--a mechanism absent from existing approaches. The literature and the investigators' pilot data indicate that patients who express emotional distress at baseline, such as high anxiety and depressive symptoms, may be particularly likely to benefit from EAET's emotion regulation approach, whereas patients who express less emotional distress may derive more benefit from an approach like CBT, which does not require ready access to emotions.

The proposed randomized clinical trial tests the hypothesis that EAET is superior to CBT on reduction in mean pain severity and other outcomes derived from IMMPACT. To examine which patients are most likely to benefit, this research also tests whether greater baseline emotional distress (using measures of anxiety and depression) predicts stronger benefits from EAET and whether lower baseline emotional distress predicts stronger benefits from CBT. Finally, this research explores whether the benefits of EAET are mediated by improved emotion regulation, whether the benefits of CBT are mediated by improved cognitive and behavioral coping, and whether the benefits of both are mediated by a stronger working alliance. These mediators (e.g., Survey of Pain Attitudes, Working Alliance Inventory) were originally listed as outcomes in the trial registration, but they have been removed. The investigators plan to enroll 160 multi-ethnic/multi-racial older Veterans (age 60-95 years) with chronic musculoskeletal pain at the West Los Angeles VA Medical Center.

This research can introduce an additional, potentially more effective format of psychotherapy at VA so that more Veterans with chronic pain can respond. In addition, this research can lead to better treatment targeting and enhance the understanding of how psychotherapy treatments work. Finally, this research can facilitate the development of critical skills for the PI in psychotherapy research and pain management and enhance his ability to effect positive change for older Veterans.

Recruitment was resumed after the COVID-19 Administrative Hold was lifted in October 2020.

ELIGIBILITY:
Inclusion Criteria:

Eligible Veterans are age 60 to 95 years old and have had at least 3 months of musculoskeletal pain, including the following conditions most likely to benefit from psychosocial intervention based on previous research:

* regional pain syndromes (e.g., low back, neck, leg, or pelvic pain, or temporomandibular joint disorders);
* widespread pain syndromes (e.g., fibromyalgia);
* whiplash;
* tension headaches; or
* any combination of these disorders.

Exclusion Criteria:

* Confirmed hip or knee osteoarthritis without other musculoskeletal pain complaints;
* Leg pain greater than back pain only without other musculoskeletal pain complaints (to exclude radiculopathy in isolation);
* EMG-confirmed "tunnel" syndromes (e.g., carpal or tarsal tunnel syndrome) only without other musculoskeletal pain complaints;
* Autoimmune disease that typically generates pain (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, ankylosing spondylitis);
* Cancer pain, sickle cell disease, neuralgias (e.g., trigeminal neuralgia), burn pain, infection associated with pain (e.g., vertebral infection), cauda equina syndrome, gout, migraine or cluster headaches without additional musculoskeletal pain complaints;
* Uncontrolled severe psychiatric disorder including current psychotic disorder or severe mood disorder not controlled with medications (e.g., schizophrenia or bipolar I disorder), dissociative identity disorder, or active suicide/violence risk in the past 6 months;
* Substantial cognitive impairment or dementia (Mini-Mental State Exam (78) score 24);
* Active severe alcohol or substance use disorder that inhibits the participant's ability to attend session or participate in homework;
* Currently with pain-related litigation or applying for pain-related compensation or compensation increase, or undergoing compensation re-evaluation (e.g., applying for VA service connection or service connection increase for pain);
* Patients who have undergone CBT for pain within the last 3 months of enrollment or who are currently receiving CBT or EAET psychotherapy treatment for pain;
* Unable to fluently read/converse in English;
* Planning to move from the area in the next 6 months.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon C Yarns, MD MS BME, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yarns BC, Jackson NJ, Alas A, Melrose RJ, Lumley MA, Sultzer DL. Emotional Awareness and Expression Therapy vs Cognitive Behavioral Therapy for Chronic Pain in Older Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2415842. doi: 10.1001/jamanetworkopen.2024.15842. PMID 38869899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics at VA Greater Los Angeles, letter-based recruitment based on a search of data from the VA Corporate Warehouse, and self-referral from flyers. The first participants was enrolled on May 16, 2019, and the last participant was enrolled on February 1, 2023. Recruitment was paused from March 20, 2020, until February 4, 2021, due to COVID-19 related administrative holds.
Pre-assignment Details: Of 126 enrolled, 126 were randomized to treatment.
Period: Overall Study
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Started | 66 | 60
Completed Posttreatment (Week 10) Assessments | 57 | 54
Completed (6-month follow-up assessments) | 54 | 50
Not Completed | 12 | 10
Not completed — Lost to Follow-up | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy | Total
Number analyzed (Participants) | 66 | 60 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (5.2) | 71.3 (6.6) | 71.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 59 | 57 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 60 | 58 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 37 | 69
  White | 22 | 17 | 39
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 6 | 2 | 8
Marital status [Count of Participants; unit: Participants]
  Married or partnered | 23 | 19 | 42
  Divorced or separated | 25 | 25 | 50
  Never married or other | 18 | 16 | 34
Education level [Count of Participants; unit: Participants]
  High school or less | 10 | 14 | 24
  Some college | 36 | 26 | 62
  College graduate or more | 20 | 20 | 40
Pain duration [Mean (Standard Deviation); unit: years] | 22.5 (18.2) | 24.4 (17.3) | 23.3 (17.7)
No. prescribed opioids at baseline [Count of Participants; unit: Participants]
  Opioids | 8 | 6 | 14
  No opioids | 58 | 54 | 112
Any psychiatric diagnosis [Count of Participants; unit: Participants]
  Psychiatric diagnosis (e.g., depression, anxiety, PTSD) | 44 | 43 | 87
  No psychiatric diagnosis | 22 | 17 | 39
VA service-connected for PTSD [Count of Participants; unit: Participants]
  VA service-connected for PTSD | 25 | 22 | 47
  Not VA service-connected for PTSD | 41 | 38 | 79
No. non-pain chronic medical conditions [Mean (Standard Deviation); unit: conditions] | 5.0 (2.2) | 4.9 (2.7) | 5.0 (2.4)
No. prescription medications [Mean (Standard Deviation); unit: medications] | 9.9 (5.2) | 9.4 (4.3) | 9.6 (4.8)
Mini-Mental State Examination Scores [Mean (Standard Deviation); unit: units on a scale] — Sum of 30 questions evaluating cognition (i.e., orientation, verbal memory registration, short-term memory recall, working memory, language, and visuospatial abilities), yielding a total score between 0 and 30 with higher scores indicating better cognition.
  units on a scale | 28.9 (1.1) | 28.4 (1.6) | 28.6 (1.4)
Back pain [Count of Participants; unit: Participants]
  Back pain | 63 | 58 | 121
  No back pain | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: Average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: Intent to Treat Population (all participants assigned to Emotional Awareness and Expression Therapy or Cognitive Behavior Therapy)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -2.18 [-3.00 to -1.37] | -0.60 [-1.13 to -0.06]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.59, 95% CI 2-sided [-2.35 to -0.83]

2. Secondary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -1.26 [-1.83 to -0.68] | -0.25 [-0.72 to 0.23]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Net) = -1.01, 95% CI 2-sided [-1.78 to -0.24]

3. Secondary Outcome: Satisfaction With Therapy and Therapist Scale-Revised (Overall Satisfaction)
Description: Overall satisfaction is a single item on the Satisfaction with Therapy and Therapist Scale-Revised scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction) with higher scores indicating a better outcome.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | 4.30 [4.05 to 4.54] | 4.01 [3.83 to 4.19]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.28, 95% CI 2-sided [0.12 to 0.45]

4. Secondary Outcome: PROMIS-Pain Interference Short Form 8a v1.0
Description: Sum of eight self-report items assessing interference of pain with daily activities over the past 7 days. Items range from 1-5 (1 = no interference; 5 = maximum interference), yielding a total score between 8 and 40 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -5.41 [-7.33 to -3.48] | -3.99 [-6.41 to -1.56]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = -1.42, 95% CI 2-sided [-3.30 to 0.46]

5. Secondary Outcome: PROMIS-Pain Interference Short Form 8a v1.0
Description: as for outcome 4
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -2.87 [-4.96 to -0.78] | -3.08 [-4.59 to -1.57]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.85, Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-1.99 to 2.42]

6. Secondary Outcome: PROMIS-Depression Short Form
Description: Sum of eight self-report items assessing depression and emotional distress over the past 7 days. Items range from 1-5 (1 = never feeling a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 8 and 40 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -5.12 [-6.62 to -3.62] | -2.06 [-4.31 to 0.20]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -3.06, 95% CI 2-sided [-5.88 to -0.25]

7. Secondary Outcome: PROMIS-Depression Short Form
Description: as for outcome 6
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -3.48 [-4.94 to -2.03] | -1.09 [-2.97 to 0.78]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -2.39, 95% CI 2-sided [-4.33 to -0.45]

8. Secondary Outcome: PROMIS-Anxiety Short Form
Description: Sum of seven self-report items assessing anxiety over the past 7 days. Items range from 1-5 (1 = never experiencing a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 7 and 35 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -3.13 [-4.56 to -1.70] | -0.64 [-2.18 to 0.89]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Net) = -2.49, 95% CI 2-sided [-4.30 to -0.68]

9. Secondary Outcome: PROMIS-Anxiety Short Form
Description: as for outcome 8
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -3.17 [-4.58 to -1.76] | -1.22 [-2.53 to 0.09]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -1.95, 95% CI 2-sided [-4.34 to 0.45]

10. Secondary Outcome: PTSD Checklist for DSM-5
Description: Sum of twenty self-report items assessing PTSD according to the frequency in which symptoms are experienced over the past month. Items range from 0-4 (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely), yielding a total score between 0 and 80 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: Intent to Treat Population (all participants assigned to Emotional Awareness and Expression Therapy or Cognitive Behavior Therapy when PTSD symptoms were assessed; groups 3-10)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 52 | 47
score on a scale | -4.45 [-7.55 to -1.34] | -0.06 [-3.55 to 3.44]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -4.39, 95% CI 2-sided [-8.44 to -0.34]

11. Secondary Outcome: PTSD Checklist for DSM-5
Description: as for outcome 10
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 52 | 47
score on a scale | -4.07 [-6.26 to -1.88] | -0.31 [-5.28 to 4.66]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -3.76, 95% CI 2-sided [-7.83 to 0.32]

12. Secondary Outcome: NIH Toolbox-Life Satisfaction Short Form
Description: Sum of five self-report items assessing general life satisfaction. Items range from 1-5 (1 = no satisfaction; 5 = maximum satisfaction), yielding a total score between 5 and 25 with higher scores indicating a better outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | 1.68 [1.02 to 2.34] | 0.45 [-0.15 to 1.05]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = 1.23, 95% CI 2-sided [0.36 to 2.10]

13. Secondary Outcome: NIH Toolbox-Life Satisfaction Short Form
Description: as for outcome 12
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | 1.15 [0.82 to 1.48] | 0.21 [-0.94 to 1.35]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Net) = 0.95, 95% CI 2-sided [-0.40 to 2.29]

14. Secondary Outcome: PROMIS-Sleep Disturbance Short Form
Description: Sum of eight self-report items assessing sleep disturbance over the past 7 days. Items range from 1-5 (1 = no sleep disturbance; 5 = maximum sleep disturbance), yielding a total score between 8 and 40 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -2.69 [-4.39 to -0.98] | -0.84 [-2.61 to 0.94]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -1.85, 95% CI 2-sided [-4.14 to 0.44]

15. Secondary Outcome: PROMIS-Sleep Disturbance Short Form
Description: as for outcome 14
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -2.73 [-4.21 to -1.24] | -0.16 [-2.21 to 1.89]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -2.57, 95% CI 2-sided [-5.73 to 0.60]

16. Secondary Outcome: PROMIS-Fatigue Short Form
Description: Sum of seven self-report items assessing fatigue over the past 7 days. Items range from 1-5 (1 = no fatigue; 5 = maximum fatigue), yielding a total score between 7 and 35 with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -1.97 [-3.00 to -0.93] | -1.19 [-2.44 to 0.06]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Net) = -0.78, 95% CI 2-sided [-2.33 to 0.78]

17. Secondary Outcome: PROMIS-Fatigue Short Form
Description: as for outcome 16
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | -1.47 [-2.53 to -0.40] | -1.17 [-2.49 to 0.15]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = -0.30, 95% CI 2-sided [-1.74 to 1.14]

18. Secondary Outcome: Patient's Global Impression of Change Scale
Description: Patient rates on a single item with a scale of 1-7 the change (if any) they've experienced since beginning treatment in the study (1 = no change or condition has worsened; 7 = a great deal better and a considerable improvement that has made all the difference) with higher scores indicating a better outcome.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | 4.67 [4.17 to 5.16] | 3.20 [2.79 to 3.61]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.46, 95% CI 2-sided [0.77 to 2.15]

19. Secondary Outcome: Patient's Global Impression of Change Scale
Description: as for outcome 18
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
score on a scale | 4.01 [3.61 to 4.41] | 2.77 [2.34 to 3.21]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.24, 95% CI 2-sided [0.62 to 1.86]

20. Secondary Outcome: Percentage of Participants With at Least 30% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10 . Mean pain severity is calculated at baseline and 10 weeks, and the two scores are compared to see if mean pain severity at 10 weeks is 30% lower than at baseline.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 63.5 [50.6 to 76.4] | 17.1 [6.8 to 27.5]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 21.54, 95% CI 2-sided [4.66 to 99.56]

21. Secondary Outcome: Percentage of Participants With at Least 30% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10. Mean pain severity is calculated at baseline and 20 weeks, and the two scores are compared to see if mean pain severity at 20 weeks is at least 30% lower than at baseline.
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 40.3 [26.8 to 53.8] | 14.2 [4.3 to 24.0]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.006, Mixed Models Analysis; Odds Ratio (OR) = 7.24, 95% CI 2-sided [1.74 to 30.06]

22. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10. Mean pain severity is calculated at baseline and 10 weeks, and the two scores are compared to see if mean pain severity at 10 weeks is at least 50% lower than at baseline.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 35.7 [21.5 to 49.8] | 7.4 [0.0 to 14.7]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.002, Mixed Models Analysis; Odds Ratio (OR) = 11.77, 95% CI 2-sided [2.38 to 58.25]

23. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10. Mean pain severity is calculated at baseline and 20 weeks, and the two scores are compared to see if mean pain severity at 20 weeks is at least 50% lower than at baseline.
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 16.6 [5.8 to 27.4] | 3.9 [0.0 to 9.4]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.05, Mixed Models Analysis; Odds Ratio (OR) = 6.58, 95% CI 2-sided [0.99 to 43.67]

24. Secondary Outcome: Percentage of Participants With at Least 70% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10. Mean pain severity is calculated at baseline and 10 weeks, and the two scores are compared to see if mean pain severity at 10 weeks is at least 70% lower than at baseline.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 12.8 [2.7 to 22.8] | 1.9 [0.0 to 5.8]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.06, Mixed Models Analysis; Odds Ratio (OR) = 13.93, 95% CI 2-sided [0.86 to 225.44]

25. Secondary Outcome: Percentage of Participants With at Least 70% Improvement in Pain Severity
Description: Mean pain severity is calculated from an average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10. Mean pain severity is calculated at baseline and 20 weeks, and the two scores are compared to see if mean pain severity at 20 weeks is at least 70% lower than at baseline.
Time Frame: Change from baseline to 20 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
Number analyzed (Participants) | 66 | 60
percentage of participants | 7.5 [0.0 to 15.3] | 2.1 [0.0 to 6.1]
Statistical Analysis 1: Comparison: Emotional Awareness and Expression Therapy vs Cognitive Behavior Therapy; Test type: Superiority; p = 0.22, Mixed Models Analysis; Odds Ratio (OR) = 5.61, 95% CI 2-sided [0.35 to 89.30]

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation, an average of 8 months.
Description: Adverse events were reported to the VA Clinical Sciences Research and Development Data Monitoring Committee and the local IRB
Arm/Group | Emotional Awareness and Expression Therapy | Cognitive Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 1/66 | 1/60
Serious Adverse Events (participants affected / at risk) | 2/66 | 1/60
Other Adverse Events (participants affected / at risk) | 10/66 | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emotional Awareness and Expression Therapy (N=66) | Cognitive Behavior Therapy (N=60)
Acute decompensated heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalized for worsening chronic rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urgent cholecystectomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emotional Awareness and Expression Therapy (N=66) | Cognitive Behavior Therapy (N=60)
Temporary worsening of pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Temporary worsening of depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03918642/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03918642/ICF_000.pdf